CLINICAL TRIAL: NCT01111903
Title: A Two Stage Trial of lénalidomide (Revlimid®) : a Phase II Study of lénalidomide as Single Agent in Asymptomatic Ovarian Cancer Patients With Increasing CA 125 in Late Relapse: Followed by a Phase I of lénalidomide in Combination With Carboplatin and Liposomal Pegylated Doxorubicin.
Brief Title: A 2 Stage Trial of Lenalidomide (REV) in Asymptomatic Ovarian Cancer Patients With Increasing CA 125 in Late Relapse
Acronym: REV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REV (GINECO-OV214)
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lenalidomide (Experimental): Phase II: lenalidomide 20 mg/day in continuous regimen. Phase I: lenalidomide 25 mg/day 21 days/28 + carboplatin AUC 5 + caelyx 30 mg/m2
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Phase II: 20 mg/day in continuous regimen Phase I: 25 mg/day 21 days/28 with carboplatine AUC 5 + caelyx 30mg/m2

SUMMARY:
Study in two stages, and with a sub-study.

DETAILED DESCRIPTION:
Stage A: To determine efficacy of lenalidomide as single agent in patients with recurrent ovarian cancer in second or third line.

Stage B: To determine the Maximum Tolerated Dose (MTD) of lenalidomide in combination with chemotherapy consisting of carboplatin and pegylated liposomal doxorubicin.

Substudy: To investigate the impact of the lenalidomide on patients' immune system affected by cancer and to look for an immunizing marker which could be predictive of the activity of the lenalidomide in the solid tumors.

ELIGIBILITY:
Inclusion Criteria:

Stage A: Patient:

* aged > 18 years.
* with a histological proven diagnosis of epithelial cancer of the ovary, the fallopian tube or extra-ovarian papillary serous tumors.
* with asymptomatic disease in progression detected by increase of CA 125 levels according to GCIG criteria during systematic follow-up, with or without measurable lesions.
* with disease in progression > 6 months after a first or second line including a platinum derivative. Patients should have received previously a taxane derivative.
* Adequate bone marrow, renal and hepatic function defined as: . WBC > 3.0 x 109/L or Neutrophils (ANC) > 1,5 x 109/L; Platelets > 100 x 109/L; Hemoglobin > 6 mmol/L (10,0 mg/dL); Bilirubin < 2 x upper normal limit of normal range; Estimated glomerular filtration rate > 50 ml/mn according to Cockroft-Gault formula.
* with ECOG performance status = 0 or 1.
* with a life expectancy of at least 16 weeks
* who have given their signed and written informed consent to participate in the trial after fully understanding the implication and constraints of the protocol.

Stage B: Patients

* aged > 18 years.
* with a histological proven diagnosis of epithelial cancer of the ovary, the fallopian tube or extra-ovarian papillary serous tumors.
* with disease in progression > 6 months after a first or second line including a platinum derivative. patients should have received previously a taxane derivative.
* Measurable disease by RECIST or evaluable disease by GCIG (CA-125).
* Patients included in stage A with disease in progression under lenalidomide could be eligible in phase B if they did not experience unacceptable toxicity under lenalidomide in stage A. Patients should stop lenalidomide for 7 days before entry in stage B (7 days wash out).
* Adequate bone marrow, renal and hepatic function defined as: . WBC > 3.0 x 109/L or Neutrophils (ANC) > 1,5 x 109/L; Platelets > 100 x 109/L; Hemoglobin > 6 mmol/L (10,0 mg/dL); Bilirubin < 2 x upper normal limit of normal range; Estimated glomerular filtration rate > 50 ml/mn according to Cockroft-Gault formula.
* with LVEF under normal range
* with ECOG performance status = 0 or 1.
* with a life expectancy of at least 16 weeks.
* who have given their signed and written informed consent to participate in the trial after fully understanding the implication and constraints of the protocol.

Exclusion Criteria:

* Ovarian tumors of low malignant potential (borderline tumors).
* Non-epithelial ovarian or mixed epithelial/non epithelial tumors (e.g. mixed Mullerian tumors).
* Patients with a prior diagnosis of any malignancy not cured by surgery alone less than 5 years before study entry (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin).
* Patients who have received previous radiotherapy.
* Presence of symptomatic brain metastases.
* Patients with a history of seizure disorder or central nervous system disorders; pre-existing motor or sensory neurologic pathology or symptoms > NCI-CTC grade 1.
* History of congestive heart failure (NYHA Classification > 2, even if medically controlled. History of clinical and electrocardiographically documented myocardial infarction within the last 6 months. History of atrial or ventricular arrhythmias (≥ LOWN II).
* Thrombosis or anti-thrombosis treatment within 6 months.
* History of visceral bleeding, gastrointestinal ulcer in 6 months.
* Obstructive or sub-occlusive disease.
* Patients with severe active infection.
* Concurrent severe medical problems unrelated to malignancy which would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy.
* Fertile women not using adequate contraceptive methods, or who are pregnant or breast feeding.
* Histories of allergy or sentimentality known about the similar chemical compounds in the carboplatine, either in the doxorubicine liposomale pégylée, or in one of the constituents of the lenalidomide.
* Patient having developed a knotty erythema characterized by a rash with desquamation during grip(taking) of thalidomide or a medicine similaire.
* Previous administration of lenalidomide.
* Seropositivity known about the virus of the human immunodeficiency (HIV), or pathology bound to the syndrome of acquired immunodeficiency (AIDS) or hepatitis activates type A, B or C.
* Administration of other simultaneous chemotherapeutic drugs, or hormonal therapy, or simultaneous radiotherapy during the study treatment period (hormone replacement therapy is allowed as are steroid antiemetics).
* Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of lenalidomide as single agent, then DMT of lenalidomise with carboplatin and pegylated liposomal doxorubicin | Rate of Tumor Response + Stable Disease (at 4 months) / DMT
  STAGE A: To determine efficacy of lenalidomide as single agent in patients with recurrent ovarian cancer in second or third line.
  STAGE B: To determine the Maximum Tolerated Dose (MTD) of lenalidomide in combination with chemotherapy consisting of carboplatin and pegylated liposomal doxorubicin.

SECONDARY OUTCOMES:
Safety profile of lenalidomide as single agent, then in combination | Response rate, Stable Disease rate at 4 months / MDT
  STAGE A:
  * To determine the safety profile of lenalidomide (type, frequency, severity, and relationship of adverse events to study treatment).
  * To assess time to progression (TTP).
  STAGE B:
  * To evaluate the safety profile of the combination therapy.
  * To determine the response rate.
  * To assess time to progression.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric SELLE, MD, Principal Investigator — Hôpital Tenon
Locations (1):
- Hopital Tenon, Paris, France

REFERENCES:
- [Derived] Selle F, Sevin E, Ray-Coquard I, Mari V, Berton-Rigaud D, Favier L, Fabbro M, Lesoin A, Lortholary A, Pujade-Lauraine E. A phase II study of lenalidomide in platinum-sensitive recurrent ovarian carcinoma. Ann Oncol. 2014 Nov;25(11):2191-2196. doi: 10.1093/annonc/mdu392. Epub 2014 Sep 10. PMID 25210017